CLINICAL TRIAL: NCT01659606
Title: Radiation- and Alkylator-free Hematopoietic Cell Transplantation for Bone Marrow Failure Due to Dyskeratosis Congenita / Telomere Disease
Brief Title: Radiation- and Alkylator-free Bone Marrow Transplantation Regimen for Patients With Dyskeratosis Congenita
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital Los Angeles (Other); Fred Hutch/University of Washington/Seattle Children's Cancer Consortium (Unknown); Baylor College of Medicine (Other); Children's Hospital of Philadelphia (Other); University of Wisconsin, Madison (Other); Karolinska University Hospital (Other); Hackensack Meridian Health (Other); Duke University (Other); Oslo University Hospital (Other); Children's Mercy Hospital Kansas City (Other); Mayo Clinic (Other); University of Chicago (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Suneet Agarwal, Associate Professor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-950; IRB-P00003466 (Other: Boston Children's Hospital)
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2025-01

CONDITIONS: Dyskeratosis Congenita; Hoyeraal Hreidarsson Syndrome; Revesz Syndrome; Aplastic Anemia
Keywords: dyskeratosis congenita; bone marrow failure; aplastic anemia; bone marrow transplantation; reduced intensity conditioning; campath; fludarabine; telomere
MeSH Terms: conditions — Dyskeratosis Congenita; Hoyeraal Hreidarsson syndrome; Revesz Debuse syndrome; Anemia, Aplastic; Bone Marrow Failure Disorders | interventions — Alemtuzumab; fludarabine; fludarabine phosphate; Cyclosporins; Cyclosporine; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- alemtuzumab/fludarabine conditioning (Experimental): alemtuzumab/fludarabine conditioning; calcineurin-inhibitor/mycophenolate mofetil GVHD prophylaxis
  Interventions: Biological: alemtuzumab; Drug: Fludarabine; Drug: Cyclosporins; Drug: Mycophenolate mofetil; Drug: Tacrolimus

INTERVENTIONS:
Biological: alemtuzumab — Conditioning: alemtuzumab 0.2 mg/kg/dose IV/SC x 5 doses
  Other Names: Campath-1H
Drug: Fludarabine — fludarabine 30 mg/m2/dose IV x 6 doses
  Other Names: Fludara
Drug: Cyclosporins
  Other Names: cyclosporine A; Neoral; Sandimmune
Drug: Mycophenolate mofetil
  Other Names: Cellcept
Drug: Tacrolimus
  Other Names: FK506; Prograf

SUMMARY:
Dyskeratosis congenita is a disease that affects numerous parts of the body, most typically causing failure of the blood system. Lung disease, liver disease and cancer are other frequent causes of illness and death. Bone marrow transplantation (BMT) can cure the blood system but can make the lung and liver disease and risk of cancer worse, because of DNA damaging agents such as alkylators and radiation that are typically used in the procedure. Based on the biology of DC, we hypothesize that it may be possible to avoid these DNA damaging agents in patients with DC, and still have a successful BMT. In this protocol we will test whether a regimen that avoids DNA alkylators and radiation can permit successful BMT without compromising survival in patients with DC.

DETAILED DESCRIPTION:
Dyskeratosis congenita (DC) is an inherited multisystem disorder, which classically presents with a clinical triad of skin pigment abnormalities, nail dystrophy, and oral leukoplakia. DC is part of a spectrum of telomere biology disorders, which include some forms of inherited idiopathic aplastic anemia, myelodysplastic syndrome, and pulmonary fibrosis and the congenital diseases Hoyeraal-Hreidarsson syndrome and Revesz syndrome. Progressive bone marrow failure (BMF) occurs in more than 80% of patients under 30 years of age and is the primary cause of morbidity and mortality, followed by pulmonary failure and malignancies. Allogeneic hematopoietic cell transplantation (HCT) is curative for the hematological defects, but several studies have demonstrated poor outcomes in DC patients due to increased early and late complications. A predisposition to pulmonary failure, vascular disease and secondary malignancies may contribute to the high incidence of fatal complications following HCT in DC patients, and provides an impetus to reduce exposure to chemotherapy and radiotherapy in preparative regimens. Recent studies suggest that fludarabine-based conditioning regimens provide stable engraftment and may avoid the toxicities seen after HCT for DC, but studies to date are limited to case reports, retrospective studies and a single prospective trial. In this study, we propose to prospectively evaluate the efficacy of a fludarabine- and antibody-based conditioning regimen in HCT for DC patients, with the goals of maintaining donor hematopoiesis and transfusion independence while decreasing early and late complications of HCT for DC.

ELIGIBILITY:
Inclusion Criteria:

* Bone marrow hypocellular for age
* Moderate or severe aplastic anemia defined by one of the following: peripheral blood neutrophils < 0.5 x 10^9/L; platelets < 30 x 10^9/L or platelet transfusion dependence; reticulocytes < 50 x 10^9/L in anemic patients or red cell transfusion dependence
* Diagnosis of dyskeratosis congenita based on clinical triad of abnormalities of skin pigmentation, nail dystrophy, oral leukoplakia; OR one of clinical triad and presence of two or more associated features; OR a pathogenic mutation in DKC1,TERC, TERT, NOP10, NHP2, TCAB1, TINF2, CTC1, PARN, RTEL1, ACD, NAF1, STN1, or ZCCHC8, as reported by a CLIA-approved laboratory; OR age-adjusted mean telomere length < 1%ile in peripheral blood lymphocytes as reported by a CLIA-approved laboratory; OR Hoyeraal-Hreidarsson syndrome; OR Revesz syndrome
* Availability of a related or unrelated donor with a 7/8 or 8/8 match for HLA-A, B, C, and DRB1.
* Patient and/or legal guardian must be able to sign informed consent.
* Donor must provide a marrow allograft.
* Diagnosis of Fanconi anemia must be excluded by mitomycin C or diepoxybutane chromosomal breakage testing on peripheral blood at a CLIA-approved laboratory (not required for patients with a genetic mutation consistent with DC)
* Adequate renal function with glomerular filtration rate equal to or greater than 30 ml/min/1.73 m2

Exclusion Criteria:

* Clonal cytogenetic abnormalities associated with MDS or AML on bone marrow examination.
* Karnofsky/Lansky performance status < 40.
* Uncontrolled bacterial, viral or fungal infections.
* Positive test for the human immunodeficiency virus (HIV).
* Pregnancy or breastfeeding.
* Known severe or life-threatening allergy or intolerance to fludarabine, alemtuzumab, mycophenolate mofetil or both cyclosporine and tacrolimus.
* Positive patient anti-donor HLA antibody, which is deemed clinically significant.
* Prior allogeneic marrow or stem cell transplantation.
* Prior solid organ transplantation.

Ages: 30 Days to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2026-07 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Primary engraftment | Up to day +100 post-BMT

SECONDARY OUTCOMES:
Survival to day+100 post-BMT | Up to day+100 post-BMT
Viral reactivation and infection | Up to day +100 post-BMT
  Number of participants with DNA virus (cytomegalovirus, Epstein Barr virus, or adenovirus) reactivation/infection detected by PCR screening will be reported.
Treatment related adverse events as assessed by CTCAE version 4.0 | Up to 1 year post-BMT
Secondary graft failure | Up to 15 years post-BMT
Acute and chronic graft-versus-host disease (GVHD) | Up to 15 years post-BMT
Engraftment monitoring (chimerism) | Up to 15 years post-BMT
Immune reconstitution as assessed by quantitation of lymphocyte subsets | Up to 15 years post-BMT
  Number of participants with quantitative defects in lymphocyte subset numbers following BMT
Changes in pulmonary function as assessed by pulmonary function testing | Up to 15 years post-BMT
Secondary malignancies | Up to 15 years post-BMT
  Number of patients with malignancies following BMT
Long-term survival | Up to 15 years post-BMT

CONTACTS AND LOCATIONS:
Overall Officials: Suneet Agarwal, MD, PHD, Principal Investigator — Boston Children's Hospital
Locations (14):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital (pediatric patients), Boston, Massachusetts
  - Dana-Farber Cancer Institute (adult patients), Boston, Massachusetts
  - Children's Mercy Hospital Kansas City, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Fred Hutch/University of Washington/Seattle Children's Cancer Consortium, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Oslo University Hospital, Oslo, Norway
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bhoopalan SV, Wlodarski M, Reiss U, Triplett B, Sharma A. Reduced-intensity conditioning-based hematopoietic cell transplantation for dyskeratosis congenita: Single-center experience and literature review. Pediatr Blood Cancer. 2021 Oct;68(10):e29177. doi: 10.1002/pbc.29177. Epub 2021 Jun 4. PMID 34086408